CLINICAL TRIAL: NCT02214602
Title: The Value of Immediate Post-operative Intravesical Epirubicin Instillation in Intermediate and High Risk Non Muscle Invasive Bladder Cancer (NMIBC): A Randomized Controlled Trial
Brief Title: Value of Immediate Post-operative Intravesical Epirubicin in Intermediate&High Risk Non Muscle Invasive Bladder Cancer
Acronym: NMIBCIVT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Resident in Urology, Urology and Nephrology Center, Mansoura University, Mansoura, Egypt, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AEl-Sawy172014
Record Dates: First submitted 2014-07-10; First posted 2014-08-12 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma of Urinary Bladder, Superficial
Keywords: non muscle invasive bladder cancer; intermediate and high risk; immediate single instillation; Intravesical chemotherapy; Disease prevention
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Epirubicin; Doxorubicin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Study group(Epirubicin) (Experimental): in this arm -study group(Epirubicin)- : patients will receive immediate intravesical instillation of 50 mg of epirubicin in 50 ml of saline 0.9 % after 30 min after compete transurethral resection of bladder tumor
  Interventions: Drug: Epirubicin
- Control group (No Intervention): in this arm -control group- : patients will not receive immediate intravesical instillation of of epirubicin after compete transurethral resection of bladder tumor.

INTERVENTIONS:
Drug: Epirubicin — Experimental: Study group(Epirubicin)
  in the arm -study group(Epirubicin)- : patients will receive immediate intravesical instillation of 50 mg of epirubicin in 50 ml of saline 0.9 % after 30 min after compete transurethral resection of bladder tumor
  Other Names: Intravesical chemotherapy; Doxorubicin
  Arms: Study group(Epirubicin)

SUMMARY:
The aim of the study is to test the value of immediate post-operative intravesical instillation of epirubicin in patients with intermediate and high risk non muscle invasive bladder cancer (NMIBC).

DETAILED DESCRIPTION:
Preoperative evaluation will be carried out in the form of routine laboratory investigations, abdominal and pelvic US and computed tomography (CT) or magnetic resonance imaging (MRI) abdomen and pelvis if necessary. Then, the patients will be subjected to complete TURBT.

The patients will be transferred to the recovery room, careful monitoring of the patients will be carried out for the 1st 30 min, and then after confirming the patient eligibility for enrollment in the study by exclusion of cases with hematuria and suspicious bladder perforation, patients will be enrolled randomly into one of the two groups. The randomization process will be performed using computer-generated simple random tables in a 1:1 ratio or by the method of closed envelopes.

The 1st group will not receive intravesical instillation of epirubicin -Placebo-(control group), and, the 2nd group will receive intravesical instillation of epirubicin 50 mg in 50 ml saline 0.9% (study group) with clamping of the urethral catheter for 1 hour after instillation and during this period the patients are monitored for local or systemic adverse events (acute abdomen, chills, fever, hot flushes, abdominal rigidity, hematuria after de-clamping of the catheter).

Evaluation:

Intraoperative and early postoperative parameters of interest will be recorded and compared between the two groups like EUA findings, tumor characteristics during cystoscopy as the tumor size, site, shape, number, suspicion of CIS, post instillation adverse events, cytology and biopsy results.

The patients will be discharged after removal of urethral catheter. They will be stratified into either intermediate or high risk histopathologically confirmed NMIBC, followed up at the outpatient clinic (OPC) and will receive adjuvant intravesical instillation of chemotherapy or immunotherapy according to the European Association of Urology (EAU) guidelines for each risk group. The patients will be evaluated by office cystoscopy and urine cytology at the OPC after 12 weeks, and thereafter every 3 months during the first 2 years and then every 3 to 6 months according to the risk category.

During the follow-up period, all histopathologically confirmed tumors will be classified as recurrences. Time to first recurrence will be the primary end point of the study, and the length of follow-up will be defined as the time from inclusion to the last cystoscopy control.

Methods of evaluation and follow-up:

All the patients will be evaluated on entry and at follow-up intervals. On study entry patients will be evaluated by urinalysis, urine culture, serum creatinine, fasting blood sugar level, complete blood count, chest X-ray, excretory urography (IVU) and or CT urography and bladder wash for cytology. CT with contrast will be performed annually in cases of high risk tumor category and when otherwise indicated. Complete TURBT of all visible tumors will be conducted in all patients and the stage and grade will be determined according to the 1987 staging classification and World Health Organization (WHO) grading system in 1973+ 2004 WHO grading system.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent.
* Patients with primary or recurrent papillary Non muscle invasive bladder cancer (NMIBC).
* Complete transurethral resection of bladder tumor(TURBT).
* Normal cardiac, hematological, and renal functions.
* Patients with intermediate and high risk NMIBC confirmed by histopathology.

Exclusion Criteria:

* Inability to give informed consent.
* Patients with history of previous radiotherapy or systemic chemotherapy.
* Patients suffering from immuno-deficiency or other malignancies.
* Patients with history of hypersensitivity reaction to epirubicin.
* Examination under anesthesia (EUA) reveals palpable bladder mass.
* Patients with primary, single, less than 1cm papillary bladder tumor (high likelihood of being low risk).
* Suspicion of perforation of the bladder during TURBT.
* Patients who develop hematuria in the recovery room necessitating continuous bladder wash or endoscopic haemostasis.
* Patients with proven low risk NMIBC on histopathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-07; Primary Completion 2017-04 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Recurrence, progression and/or death from cancer. | within the 1st year after complete Transurethral resection of bladder tumor

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | within 1st 24 hours following intravesical instillation of the used drug

CONTACTS AND LOCATIONS:
Overall Officials: Bedeir A El-Dein, Professor, Study Chair — Urology And Nephrology Center, Mansoura University, Mansoura
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Egypt

REFERENCES:
- [Derived] Elsawy AA, El-Assmy AM, Bazeed MA, Ali-El-Dein B. The value of immediate postoperative intravesical epirubicin instillation as an adjunct to standard adjuvant treatment in intermediate and high-risk non-muscle-invasive bladder cancer: A preliminary results of randomized controlled trial. Urol Oncol. 2019 Mar;37(3):179.e9-179.e18. doi: 10.1016/j.urolonc.2018.10.019. Epub 2018 Nov 14. PMID 30448030